CLINICAL TRIAL: NCT01084161
Title: A Randomized Double-Blind, Placebo- and Active-Controlled, Dose-Ranging Study to Evaluate the Analgesic, Efficacy, Safety and Tolerability of Intravenous N1539 in Subjects After Open Abdominal Hysterectomy
Brief Title: Study to Evaluate the Efficacy, Safety and Tolerability of N1539
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: N1539-04
Record Dates: First submitted 2010-03-05; First posted 2010-03-10 (Estimated); Last update posted 2011-12-02 (Estimated); Status verified 2011-11

CONDITIONS: Hysterectomy
MeSH Terms: interventions — Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (7):
- N1539 5 mg (Experimental)
  Interventions: Drug: N1539
- N1539 7.5 mg (Experimental)
  Interventions: Drug: N1539
- N1539 15 mg (Experimental)
  Interventions: Drug: N1539
- N1539 30 mg (Experimental)
  Interventions: Drug: N1539
- N1539 60 mg (Experimental)
  Interventions: Drug: N1539
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo
- morphine (Active Comparator)
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: N1539 — 5 mg IV once per day
  Arms: N1539 5 mg
Drug: N1539 — 7.5 mg IV once per day
  Arms: N1539 7.5 mg
Drug: N1539 — 15 mg IV once per day
  Arms: N1539 15 mg
Drug: N1539 — 30 mg IV once per day
  Arms: N1539 30 mg
Drug: placebo — IV placebo once per day
  Arms: Placebo
Drug: Morphine — morphine 10-15 mg IV once per day
  Arms: morphine
Drug: N1539 — 60 mg IV once per day
  Arms: N1539 60 mg

SUMMARY:
To determine the analgesic efficacy, duration of effect, and safety of single doses of N1539 in subjects undergoing open abdominal hysterectomy

ELIGIBILITY:
Inclusion Criteria:

* moderate to severe pain with VAS of >/= 45 mm
* undergo open abdominal hysterectomy
* ASA I or II
* signed ICF
* BMI >18.5 and < 31.5 kg/m^2

Exclusion Criteria:

* suspected metastatic cervical or endometrial cancer
* prior abdominal surgery with postoperative complications
* active pancreatitis, obstruction of biliary tree or total bilirubin> 2.5 mg/dL
* active GI bleeding, or peptic ulcer disease
* unstable medical condition
* HbA1c >9.5 or uncontrolled diabetes
* SBP >150 mmHg or DBP > 95 mmHg
* personal or familial contraindication to undergoing general anesthesia
* Antihypertensive agents or diabetic regimen that is not stable (4 weeks prior to surgery)
* taking CNS agents for pain
* acetaminophen or NSAIDs not discontinued for at least 5 half-lives prior to planned surgery
* currently taking an opioid or has taken an opioid chronically for pain in past 2 years
* corticosteroid or systemic corticosteroids within 6 weeks of planned surgery
* has a known bleeding disorder or taking agents affecting coagulation
* history of intolerance or allergic reactions to NSAIDs, COX-2 inhibitors, aspirin and other salicylates
* receiving lithium or a combination of furosemide with an ACE inhibitor or angiotensin receptor blocker
* Known to have sleep apnea
* History of hepatitis B or C
* AST or ALT > 2 times the upper limit of normal
* Known or suspected COPD with retention of carbon dioxide
* psychiatric condition that impairs the capability of the subject to report pain

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 486 (Actual)
Dates: Start 2010-03; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
To determine the analgesic efficacy, duration of effect and safety of single doses of IV N1539 as measured by the SPID (summary of pain intensity) and TOPAR (summary of the time-weighted pain relief scores) from 0-24 hours. | at 60 minutes post dose and at 24 hours
  Additionally, to determine the efficacy seen within the first hour after study drug administration, as measured by the SPID 0-60 minutes post-dose.

SECONDARY OUTCOMES:
To assess the safety and tolerability of IV N1539 by laboratory data, vital signs, wound site evaluation and Adverse Events | 5-7 days post initial dosing

CONTACTS AND LOCATIONS:
Locations (11):
- Tbilisi, Georgia
- Poland (7):
  - Bialystok
  - Gdansk
  - Lodz
  - Lublin
  - Poznan
  - Ruda Śląska
  - Szczecin
- Serbia (3):
  - Belgrade
  - Kragujevac
  - Novi Sad

REFERENCES:
- [Derived] Rechberger T, Mack RJ, McCallum SW, Du W, Freyer A. Analgesic Efficacy and Safety of Intravenous Meloxicam in Subjects With Moderate-to-Severe Pain After Open Abdominal Hysterectomy: A Phase 2 Randomized Clinical Trial. Anesth Analg. 2019 Jun;128(6):1309-1318. doi: 10.1213/ANE.0000000000003920. PMID 31094806
- [Derived] Viscusi ER, Gan TJ, Bergese S, Singla N, Mack RJ, McCallum SW, Du W, Hobson S. Intravenous meloxicam for the treatment of moderate to severe acute pain: a pooled analysis of safety and opioid-reducing effects. Reg Anesth Pain Med. 2019 Mar;44(3):360-368. doi: 10.1136/rapm-2018-100184. Epub 2019 Feb 7. PMID 30737315